CLINICAL TRIAL: NCT03647748
Title: Effects of Green Light Therapy on Body Contouring and Cellulite
Acronym: Cellulize
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ward Photonics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CP16-02
Record Dates: First submitted 2018-08-20; First posted 2018-08-27 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Fat Reduction

STUDY DESIGN:
Intervention Model Description: Patients randomly assigned to either the active 532nm treatment group, or the sham device (placebo) group using a modified device rigged to not treat patients.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cellulize 532nm (No Intervention): Cellulize device using 532nm Green Light.
- Cellulize Placebo (Sham Comparator) (Sham Comparator): Cellulize modified to appear as if it is running, but does not use the 532nm light.
  "Sham" Device, or "Placebo."
  Interventions: Device: Sham Comparator

INTERVENTIONS:
Device: Sham Comparator — A modified device utilizing a pigtail connector to bypass active treatment.
  Arms: Cellulize Placebo (Sham Comparator)

SUMMARY:
A double-blind, placebo-controlled randomized evaluation of the effect of Cellulize, a green light low level laser system for aesthetic use for the non-invasive reduction in fat layer for body contouring and reduction of cellulite.

DETAILED DESCRIPTION:
This clinical trial will provide objective evidence showing effectiveness of the Cellulize 532nm green light therapy for the non-invasive reduction in fat layer for body contouring, and for the non-invasive treatment for the appearance of cellulite.

ELIGIBILITY:
Inclusion Criteria:

* Study participant between the ages of 18 and older.
* Female only
* Subject is willing and able to abstain from partaking in any treatment other than the study procedures (existing or new) to promote body contouring/circumference reduction/weight loss during the course of study participation.
* Subject is willing and able to maintain his or her regular (typical pre-study) diet and exercise regimen without effecting significant change in either direction during study participation.

Exclusion Criteria:

* No photo-therapy (red or green) within 3 weeks of treatment.
* Known cardiovascular disease such as cardiac arrhythmias, congestive heart failure.
* Cardiac surgeries such as cardiac bypass, heart transplant surgery, pacemakers.
* Prior surgical intervention for body sculpting/weight loss, such as liposuction, abdominoplasty, stomach stapling, lap band surgery, etc.
* Medical, physical, or other contraindications for body sculpting/weight loss.
* Current use of medication(s) known to affect weight levels/cause bloating or swelling and for which abstinence during the course of study participation is not safe or medically prudent.
* Any medical condition known to affect weight levels and/or to cause bloating or swelling.
* Active infection, open wound (e.g. sores, cuts, ulcers, burns, etc.) or other external trauma to the areas to be treated with the laser/lymphatic drainage system devices.
* Photosensitive condition or medication.
* Active cancer within the past year.
* Pregnant, possibly pregnant or planning pregnancy prior to the end of study participation.
* Diminished ability to void waste (liver or kidneys).
* Developmental disability or cognitive impairment that in the opinion of the investigator would preclude adequate comprehension of the informed consent form and/or ability to record the necessary study measurements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Average Change in Inches of Total Circumference Measurements | 2 weeks
  Average Change in Inches of Total Circumference Measurements for effect of Cellulize, a LED 532nm green light low level laser system for aesthetic use for the non-invasive reduction in fat layer for body contouring from baseline measurements, and after treatment.

SECONDARY OUTCOMES:
Durability of Effect | 2 weeks
  Durability of Effect: a term used to indicate whether the results of the primary outcome endure at the 2 week follow up time point. If the average change in inches of total circumference continues decreasing or stays the same, then the durability of effect is assumed to endure for at least two weeks. If the measurements at the 2-week time point show that the changes in inches return to previous measures at the start of treatment, then the effect is considered temporary.
Change in appearance of cellulite | 2 weeks
  Change in appearance of cellulite is a measure of the Nurnberger-Muller Scale (NMS) from baseline to 2 weeks post-assessment for both of the right and left thighs.

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Burke, MD, Study Director — Michigan Center for Cosmetic Surgery, Ann Arbor, Michigan
Locations (4):
- United States (4):
  - Wunderlich Chiropractic Clinic, Cape Coral, Florida
  - Mobile Laser Slimming, Cocoa Beach, Florida
  - Lake Mary Health and Wellness, Lake Mary, Florida
  - Michigan Center for Cosmetic Surgery, Ann Arbor, Michigan, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No